

# **RESEARCH PARTICIPANT INFORMED CONSENT FORM**(WEB-BASED PILOT TEST)

Please read this document carefully before you decide to participate in this research study. Your participation is voluntary, and you can decline to participate, or withdraw consent at any time, with no consequences.

#### **Study Title:**

Adapting and Pilot Testing a Nutrition Module delivered with Virtual Human Technology for Colorectal Cancer Prevention

#### Person(s) conducting the research:

Melissa Vilaro, Postdoctoral Associate, STEM Translational Communication Center, College of Journalism and Communications, University of Florida, <a href="mailto:mgraveley@ufl.edu">mgraveley@ufl.edu</a>, (352) 846-3014

Janice Krieger, Director, STEM Translational Communication Center, College of Journalism and Communications, University of Florida, <u>Janicekrieger@ufl.edu</u>, (352) 273-0204

Ben Lok, Professor, Computer & Information Sciences & Engineering Department, University of Florida, <a href="mailto:lok@cise.ufl.edu">lok@cise.ufl.edu</a>, (352) 450-6308

# Purpose of the research study:

This study uses the opinions of adults between the ages of 45 and 73 years old to develop and test an interactive nutrition module for use in an existing colorectal cancer screening intervention using virtual human technology. This study will contribute to knowledge of what messages and graphics promote understanding of cancer risk and promote screening.

## What you will be asked to do in the study:

You will be asked to interact with an interactive web-based application (or app) containing a virtual health assistant that will talk to you about nutrition and colorectal cancer screening. Directly after interacting with the virtual health assistant, you will be asked to answer a questionnaire about your demographic characteristics (ex. marital status, race, gender), health behaviors, and experiences with the virtual human app.

IRB Project #: IRB201902537 

IRB Version: 2/15/2022

PI Version: 3/19/2024 1:33 PM

#### Time required:

Approximately 25 minutes.

#### Risks and benefits:

There are no risks or discomforts anticipated. There are no direct benefits of participation for you. As a result of participation in the study, you may have a better understanding of your health.

#### **Confidentiality:**

Your identity will be kept confidential to the extent provided by law. Researchers will take every precaution to maintain confidentiality of the information you share. Information will be kept on a password protected computer and/or an encrypted hard drive. Your name will not be used in any report.

Only the researchers will have access to the information we collect online. There is a minimal risk that security of any online data may be breached, but since no identifying information will be collected, and the online host (Qualtrics) uses several forms of encryption other protections, it is unlikely that a security breach of the online data will result in any adverse consequence for you.

## **Compensation:**

Qualtrics panel participants will be compensated using the Qualtrics platform.

# Source(s) of funding for the research:

Funding for this study is provided by National Institutes of Health (NIH) National Cancer Institute (NCI) as a supplement under award number R01CA207689-02.

# May the researcher(s) benefit from the research?

We may benefit professionally if the results of the study are presented at meetings or in scientific journals.

# Withdrawal from the study:

IRB Project #: IRB201902537


IRB Version: 2/15/2022

PI Version: 3/19/2024 1:33 PM

You are free to withdraw your consent and to stop participating in this study at any time without consequence. You can decline to answer any question you don't wish to answer.

#### If you withdraw, will your information be used or discarded?

Information collected will be used up until the withdrawn date/time, unless the participant requests for the data collected to not be used.

If you wish to discuss the information above or any discomforts you may experience, please ask questions now or contact one of the research team members listed at the top of this form.

If you have any questions regarding your rights as a research subject, please contact the Institutional Review Board (IRB02) office (University of Florida; PO Box 100173; Gainesville, FL 32610; (352) 392-0433 or irb2@ufl.edu.)

## **Agreement:**

Now that you've read about the study, if you wish to participate, click the "I agree to participate" button to continue; if you do not consent to participate, click "I do not wish to participate" or just close this window.

- I agree to participate
- I do not wish to participate

IRB Project #: IRB201902537 

IRB Version: 2/15/2022

PI Version: 3/19/2024 1:33 PM